CLINICAL TRIAL: NCT02750995
Title: Peptide Vaccination in Combination With Azacitidine for Patients With Myelodysplastic Syndrome and Acute Myeloid Leukemia - A Phase I Study
Brief Title: Peptide Vaccination in Combination With Azacitidine for Patients With MDS and AML
Acronym: AZACTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel El Fassi (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Sponsor-Investigator, Daniel El Fassi, Clinical Associate Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZACTA
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: myelodysplastic syndrome; acute myeloid leukemia; azacitidine; peptide vaccine; cancer testis antigen; cancer vaccine; immunotherapy; combination therapy; NY-ESO-1; PRAME; MAGE-A3; WT-1; vaccine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination (Experimental): Azacitidine + NPMW-peptide vaccine
  Interventions: Biological: NPMW-peptide vaccine; Drug: Azacitidine

INTERVENTIONS:
Biological: NPMW-peptide vaccine — Peptide vaccine against long peptide sequences from NY-ESO-1, PRAME, MAGE-A3, WT-1.
Drug: Azacitidine — Standard therapy. All participants receive azacitidine 6 months prior to inclusion, which continues during the study period.
  Other Names: Vidaza

SUMMARY:
The purpose of this phase I study is to investigate the combination of hypomethylating agents with experimental peptide vaccination against four selected tumor antigens, known to be upregulated in response to hypomethylating agents, in patients with high risk myelodysplastic syndrome and acute myeloid leukemia.

DETAILED DESCRIPTION:
INTRODUCTION

Patients with high-risk myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML), who cannot be offered curative treatment, have a poor prognosis with a median survival of 11.5 months. There is currently only one registered drug that has been shown to prolong survival in this patient group; the hypomethylating agent azacitidine (also known as 5-azacytidine or Vidaza®). The treatment is not curative, but increases the median survival to approximately two years. The dominant cause of death is progressive disease, and there is a huge need for new treatment options.

In this study we will combine experimental immunotherapy of peptide vaccination with standard therapy of azacitidine for treatment of patients with high-risk myelodysplastic syndrome or acute myeloid leukemia. Our project is expected to expand the knowledge in regard to combination of immunotherapy and conventional treatment and will be essential for further development of this treatment modality.

MYELODYSPLASTIC SYNDROME (MDS)

Accumulation of both genetic and epigenetic changes in hematopoietic stem cells is considered the background for development of MDS. In the early stages of the disease, there is increased apoptosis, but as the disease progresses to high-risk MDS or AML there is an accumulation of chromosomal breakage, point mutations and promoter hypermethylation of tumor suppressor genes, resulting in a more aggressive and proliferative disease. The clinical symptoms are anemia, repeated infections and bleeding episodes associated with the dysfunctional bone marrow.

Currently, the only curative treatment option for MDS is allogeneic bone marrow transplantation. This is a high-risk treatment, only feasible in younger patients with a suitable donor. In 2009, a Phase III study (AZA 001) was published, showing that patients with high-risk MDS and AML with <30% blasts treated with the hypomethylating drug azacitidine had superior overall survival.

AZACITIDINE

The effect of azacitidine is not immediate in all patients, and it is therefore necessary to proceed with a minimum 5-6 cycles to determine whether the patient has a response to treatment. At present, azacitidine is the standard of care for all patients with high-risk MDS and AML with <30% blasts, who cannot be offered curative treatment. Unfortunately, most patients who respond to treatment later relapse and die of their disease. The mechanism behind the clinical efficacy of azacitidine is not fully elucidated and may be multiparametric. The hypomethylation results in re-expression of tumor suppressor genes that may serve as a possible mechanism for growth arrest. In addition, an up-regulation of cancer testis antigens (CTA) has been observed during treatment, which could lead to increased immune recognition of tumor cells, and hence immune-mediated tumor cell killing.

For participants in this trial, azacitidine is standard therapy and will be administered according to standard dosing regimens, and participants will be evaluated for treatment response according to standard criteria.

TUMOR ASSOCIATED ANTIGENS

The principle behind cancer vaccination is based on the immune system's ability to discriminate between normal and malignant cells. The immune system recognizes an altered pattern of peptide expression on the surface of the malignant cells. The altered pattern may involve the expression of qualitatively altered cell proteins, simple overexpression of normally occurring proteins, or de novo expression of proteins/glycoproteins not normally expressed in that tissue. This category of immune-recognized proteins is known as tumor associated antigens. As proteins are degraded in cells, peptides are presented on the surface of these cells as a complex with tissue type molecules (HLA molecules). T-cells may then recognize the peptide-HLA complexes, via its T-cell receptor, potentially resulting in tumor-cell killing, if sufficient priming takes place.

For the present study, the group of cancer testis antigens (CTA's) are of special interest, since expression of these are known to be regulated by methylation, and therefore affected by hypo-methylating treatment such as azacitidine. CTA's are known to be immunogenic and are only expressed at immunoprivileged sites, thus out of reach of immune responses, and on cancer cells, making them ideal targets for therapeutic cancer vaccination.

VACCINE DESIGN

We have chosen specifically three CTA's for which abundant re-expression has been shown following azacitidine treatment, including NY-ESO-1, MAGE-A3 and PRAME. WT-1 is additionally included as this protein has proven to be an important antigen in hematological malignancies and is likewise upregulated in response to azacitidine treatment.

The peptides we have chosen have not been used together in this particular combination before, but separately their use as therapeutic vaccination is well studied. Both smaller peptide sequences and full length proteins have been utilized.

The use of synthetic long peptides for induction and T-cell responses has shown superior effects in contrast to minimal peptide sequences in both mice and humans, furthermore synthetic long peptide has been shown to be efficiently processed and presented to both CD4 and CD8 T-cells of the immune system. Also, long-peptides have the advantage to enable presentation of several different T-cell epitopes dependent on the patients' HLA type. Thus, the choice of long peptides will minimize the impact of patients HLA type, and therefore in the present study allow inclusion of participants without prior selection based on HLA expression.

The peptides we have chosen are between 25 and 29 amino acids and will be mixed as a suspension with Montanide ISA-51; a commonly used water and oil based vaccine adjuvant, involved in over 150 registered trials at Clinicaltrail.gov.

TRIAL DESIGN

Patients with high-risk MDS and AML with <30% blasts are today offered treatment with azacitidine, 100 mg/m2 for 5 days every 4th week. In the proposed vaccination protocol, we have chosen to follow this same regimen, but in addition offer vaccination with peptides derived for cancer testis antigens. Patients will be included after completion of 6 courses of azacitidine and a treatment evaluation. If the patient shows response to treatment with azacitidine and the marrow is not hypoplastic, azacitidine treatment will be combined with peptide vaccination to boost the immune reactivity against selected tumor antigens. Patients will be vaccinated with a set of 3 vaccinations, with a vaccination on the 1st day of each azacitidine course, given every 4th week. If treatment is delayed more than 3 weeks the patient is excluded from the protocol. Patients are evaluated for clinical responses after 6 courses of azacitidine treatment combined with vaccination. Patients that are not progressing, will continue azacitidine treatment according to standard schedule, and further vaccinations will be given once every 6th month. Vaccination is continued for up to 2 years after initiation of vaccination or until disease progression.

STUDY METHOD

PREPARATION OF THE PEPTIDE VACCINE

The peptide vaccine will be prepared under GMP approved laboratory conditions (approved by the Danish Medicines Agency), which assures the quality of a sterile medicinal product. Production takes place in room JM702, Herlev Hospital under the approval number 24223.

Below is a brief description of the various procedures. The final vaccine product will hold a label providing information about the vaccine content and the project number given by the department.

Peptides

The vaccination will be targeted against four long peptide sequences from the proteins:

NY-ESO-1 (119-143, 25aa): PGVLLKEFTVSGNILTIRLTAADHR ; PRAME (423-447, 25aa): LQSLLQHLIGLSNLTHVLYPVPLES ; MAGE-A3 (255-279, 25aa): YLEYRQVPGSDPACYEFLWGPRALV ; WT1 (231-259, 29aa): SQLECMTWNQMNLGATLKGVAAGSSSSVK.

The peptides will be synthesized to >97% purity by an external provider, Pepscan Presto, The Netherlands. Prior to use, it will be dissolved in DMSO, mixed, and sterile filtered through a 0.22 micron filter. Endotoxin and bacterial cultivation tests will be carried out on the preparations. Sterility tests before release of peptides for vaccination treatment is carried out by hematological laboratory (location 54P4).

Adjuvant: Montanide ISA 51

Montanide ISA 51 is purchased from Seppic Inc., France, in sterile form. We will use 0.5 ml of Montanide per vaccine.

Preparation of vaccine

The vaccine will be generated as a mix of the peptide-preparation and the adjuvant, on-side, just prior to injection.

Microbiological control

Before use, the peptide mix is subjected to endotoxin tests and microbiological tests executed by the Department of Microbiology, Herlev Hospital.

EXPERIMENTAL DESIGN

This is an open-label Phase I study designed to evaluate the safety of combination therapy of azacitidine and peptide-vaccination in patients with MDS or AML.

We expect to enroll all participants within 24 months and evaluate the study 12 months thereafter. Participants will continue with azacitidine until disease progression, and with vaccination for up to 2 years, or until disease progression. Participants may stop treatment at any time upon their own request, or will be withdrawn from treatment following disease progression or severe toxicity during treatment. The inclusion period is expected to begin in April 2016 and to be finalized in April 2018. Thereafter a follow-up period of maximum 2 years is following. Last participant last protocolled visit date will be at latest, April 2020.

Patients with MDS and AML, who receive treatment with azacitidine, will be recruited through the Department of Hematology at Herlev Hospital. Since all patients are followed in an outpatient setting, for around six months prior to inclusion while receiving azacitidine treatment, possible candidates can be identified early and properly informed before a consent form needs to be signed.

ETHICAL ASPECTS

Participation is voluntary and is preceded by written informed consent. Treatment will be terminated in cases of unacceptable side effects, or upon patient's request at any time. If a patient is not interested in participation in the trial, treatment will be given according to the department's usual guidelines. The study is therefore considered ethically sound.

The study follows the guidelines of the Helsinki Agreement and the responsible physician obtains a permit from the Scientific Ethical Committee, the Danish Health and Medicines Agency and the Danish Data Protection Agency to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have received 6 courses of azacitidine and been evaluated with response to treatment.
2. Histologically confirmed high-risk MDS or AML (<30% blasts) and a normo- or hypercellular marrow after 6 courses of azacitidine.
3. Indication for continued treatment with azacitidine.
4. Age >18 years.
5. Signed consent form after receiving both written and oral information.
6. The patients must be willing to follow the scheduled treatment and sampling.

Exclusion Criteria:

1. Hypocellular bone marrow after 6 courses of azacitidine.
2. Additional active cancer disease. Participants treated for a second malignancy may be included if the patient is without evidence of disease at least 2 years after completion of treatment.
3. Participants with a known hypersensitivity to any of the active substances or to any of the excipients.
4. Participants with secondary MDS or AML
5. Severe allergies or previous anaphylactic reactions.
6. Active autoimmune disease, for example autoimmune neutropenia/ thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, Sjögren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, Addison's disease, Hashimoto's thyroiditis, Grave's disease.
7. Concomitant treatment with systemic immunosuppressive medications (including prednisone, methotrexate etc.). Participants are allowed to receive up to 10 mg prednisone at the days of azacitidine injection.
8. Concomitant treatment with other experimental drugs.
9. Concomitant treatment with other systemic anti-cancer therapy.
10. Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, up to 24 months.
  The safety of combining azacitidine treatment with this peptide vaccine will be judged on basis of the reported adverse events during the study period.

SECONDARY OUTCOMES:
Immunological evaluation | weeks: 0, 1, 9, 21. Thereafter months: 12, 18, 24
  Measurements of specific T-cell reactivity against the vaccine components. The immunological response observed before, during and after treatment will be evaluated and compared. Analyses will be performed both on blood and bone marrow samples.

OTHER OUTCOMES:
Clinical efficacy | Months: 6, 12, 18, 24
  The clinical efficacy of the treatment will be judged by the objective response rate according to the IWG modified response criteria, transfusion requirements and time to progression and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel El Fassi, MD PhD, Principal Investigator — Herlev Hospital
Locations (1):
- Dept of Hematology, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary, secondary and tertiary outcome measurements will be made available within 6 months of study completion.